CLINICAL TRIAL: NCT04401813
Title: An Open-label, Single-arm, Phase Ib Study of the Efficacy and Safety of IBI310 Combined with Sintilimab in Patients with Advanced Hepatocellular Carcinoma
Brief Title: Efficacy and Safety of IBI310 Combined with Sintilimab in Patients with Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI310C101
Record Dates: First submitted 2020-05-06; First posted 2020-05-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Advanced Hepatocellular Carcinoma
MeSH Terms: interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IBI310 (Experimental): An open-label, single-arm, Ib study of the efficacy and safety of IBI310 combined with sintilimab in patients with advanced hepatocellular carcinoma
  Interventions: Drug: IBI308 200mg

INTERVENTIONS:
Drug: IBI308 200mg — Received IBI310 combined with sintilizumab 200mg

SUMMARY:
An open-label, single-arm, Ib study of the efficacy and safety of IBI310 combined with sintilimab in patients with advanced hepatocellular carcinoma

DETAILED DESCRIPTION:
In this study, approximately 18 to 47 patients who have previously received sorafenib, lenvatinib, or oxaliplatin-containing chemotherapy . After determining the dose of IBI310, the study will enter the expansion phase

ELIGIBILITY:
inclusion criteria：

1. Locally advanced or metastatic hepatocellular carcinoma, confirmed by histology/cytology.
2. Disease progression after surgery and / or local treatment.
3. Previous standard systemic treatments for advanced hepatocellular carcinoma have failed or developed intolerable toxicity.

exclusion criteria：

1. Histology contains fibrous lamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, cholangiocarcinoma and other components.
2. Have a history of hepatic encephalopathy, or have a history of liver transplantation.
3. Diffuse liver cancer.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
adverse event | 21-42days
Evaluation of the objective response rate of IBI310 combined with 308 in the second-line treatment of advanced hepatocellular carcinoma | 21-42days

SECONDARY OUTCOMES:
Evaluate the ORR of IBI310 combined with 308 in the second-line treatment of advanced hepatocellular carcinoma (researched by the investigator according to RECIST V1.1). | 1years

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No